CLINICAL TRIAL: NCT06818110
Title: The Feasibility, Safety and Tolerability of an Exercise Training Programme in Patients with Severe Aortic Stenosis Prior to Aortic Valve Replacement Surgery: a Feasibility Trial
Brief Title: The CardioFit Trial: Exercise Training Before Aortic Valve Surgery
Acronym: CardioFit
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RHM CAR0655
Record Dates: First submitted 2024-11-27; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-11

CONDITIONS: Aortic Stenosis, Severe
Keywords: Exercise; Prehabilitation; Aortic valve replacement; Aortic stenosis; Cardiac surgery
MeSH Terms: conditions — Aortic Valve Stenosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- An in-hospital Structured Responsive Exercise-Training Programme (SRETP) (Other): Participants will participate in a structured, responsive, exercise training programme (SRETP) on a cycle ergometer. This training programme has been used in numerous international clinical trials, in several patient cohorts including cancer and lung disease.
  The training programme will involve short periods of exercise at a high intensity interspersed with short periods of exercise at a moderate intensity. This mode of exercise training is termed aerobic high-intensity interval training (HIIT). Exercise intensities during the interval exercise training program are specific to each participant and will be derived from the CPET. Moderate-intensity exercise is recognised as exercise below the anaerobic threshold. Participants will exercise at 80% of the work rate achieved at the anaerobic threshold (80%AT) for moderate-intensity exercise. High-intensity exercise is recognised as 50% of the difference between the "V" ̇O2 at the anaerobic threshold and the "V" ̇O2 peak (50%∆).
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The supervised exercise-training sessions will last <1 hour, and exercise-training intensities will be individually tailored to each participant using the results from their CPET. Participants will be screened prior to each session to ensure that it is safe to perform exercise. Exercise training will involve repeated exercise bouts of 3 minutes at a moderate exercise intensity (80%AT) followed by 2 minutes of exercise at a high-intensity (50%∆) for a predetermined amount of time. Five minutes of freewheel cycling will be performed at the start and end of the protocol for a warm-up and cool-down. Exercise sessions can be terminated by the participant at any time. Participants will have continuous ECG and SpO2 monitoring throughout the training session. Vital signs will be taken before (some during) and after each training session.
  Other Names: An in-hospital Structured Responsive Exercise-Training Programme (SRETP)

SUMMARY:
The CardioFit Trial: The feasibility, safety and tolerability of an exercise training programme in patients with severe aortic stenosis prior to aortic valve replacement surgery: A feasibility trial To investigate if a Structured Responsive Exercise Training Programme (SRETP) delivered before aortic valve replacement (AVR) in patients with severe aortic stenosis is feasible, safe, and tolerable.

Fitter patients have better surgical outcomes. Exercising post AVR surgery has been well documented and supported through cardiac rehabilitation programmes. However, there is limited evidence investigating exercising patients preoperatively, in part related to safety considerations in patients with severe aortic stenosis. If undertaking a SRETP before AVR in patients with severe aortic stenosis is shown to be feasible and safe, it provides a prehabilitation opportunity to enhance physical fitness with the aim of improving surgical outcomes.

Therefore, this trial will investigate whether SRETP (Prehabilitation) delivered before AVR in patients with severe aortic stenosis is safe & feasible.

DETAILED DESCRIPTION:
Single-centre Feasibility trial 15 patients

* Age ≥ 18 years old
* Severe aortic stenosis with a multidisciplinary team (MDT) plan for elective, aortic valve replacement
* At least 14 days until planned to come in (TCI) date
* Diagnosis of critical aortic stenosis defined as a mean gradient of ≥60mmHg or Vmax ≥5 m/s
* Presyncope/syncope due to aortic stenosis
* Unstable angina/indication for urgent surgery
* Malignant arrhythmias
* Known pregnancy
* Patients declining surgery
* Patients weight exceeds 160kg
* Patients unable to give informed consent

Intervention: 1) An in-hospital Structured Responsive Exercise-Training Programme (SRETP). The intervention will be delivered before surgery.

Feasibility Outcomes:

1. Adherence to the intervention of ≥75%
2. Tolerability of the intervention (minutes completed during the interval training) of ≥75%
3. Adverse Events to SRETP

   * Currently participating in another interventional clinical trial (this will be reviewed on a case-by-case basis)

Contraindications to SRETP:

* Acute systemic illness or fever
* Uncontrolled atrial or ventricular arrhythmias
* Uncontrolled sinus tachycardia (heart rate >120bpm)
* Acute pericarditis or myocarditis
* Decompensated heart failure
* Second or Third degree (complete) atrioventricular block without pacemaker
* Recent pulmonary embolism or deep vein thrombosis within 2 weeks
* Patients are unable to perform CPET (e.g. severe musculoskeletal conditions)

ELIGIBILITY:
Inclusion Criteria: 4.1. INCLUSION CRITERIA

Participants may enter the study if ALL of the following apply:

* Age ≥ 18 years old
* Severe aortic stenosis with a multidisciplinary team (MDT) plan for elective, aortic valve replacement
* At least 14 days until planned to come in (TCI) date.

Exclusion Criteria:4.2. EXCLUSION CRITERIA

* Diagnosis of critical aortic stenosis defined as a mean gradient of ≥60mmHg or Vmax ≥5 m/s
* Presyncope/syncope due to aortic stenosis
* Unstable angina/indication for urgent surgery
* Malignant arrhythmias
* Known pregnancy
* Patients declining surgery
* Patients weight exceeds 160kg
* Patients unable to give informed consent
* Currently participating in another interventional clinical trial (although this will be reviewed on a case-by-case basis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility Outcomes | Baseline up to surgery
  1. Adherence to the intervention ≥75%
  2. Tolerability of the intervention (minutes completed during the interval training) of ≥75%
  3. Adverse Events to the intervention (defined as occurring during or up to 30-minutes post exercise training)

SECONDARY OUTCOMES:
Endurance time | Baseline up to surgery
  Change in time to limit of tolerance (endurance time) as measured by a constant work-rate exercise test
Change in objectively measured cardiopulmonary exercise testing variables | Baseline up to surgery
  Measure a change in cardiopulmonary exercise variables. These include but are not limited to:
  Oxygen uptake (VO2) at anaerobic threshold (AT)
  Oxygen uptake at peak exercise
  VE/VCO2 slope
  Oxygen pulse
Health-related quality of life | Baseline up to surgery
  Changes in health related quality of life measurements using validated questionnaires including:
  EQ-5D-5L: A standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal
  Toronto Aortic Stenosis Quality of Life Questionnaire (TASQ-Q): A validated, brief, self-administered tool to measure changes in quality of life in patients with aortic stenosis undergoing an intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hopsitals Southampton NHS FT, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in sickle cell anemia. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: "Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis."
Access Criteria: Completion of trial